CLINICAL TRIAL: NCT00158262
Title: Prophylaxis of Posttraumatic Stress Disorder With Post-Trauma Propranolol
Brief Title: Effect of Propranolol on Preventing Posttraumatic Stress Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Roger K. Pitman, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R01MH068603 (NIH); R01MH068603 (NIH)
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Results first posted 2017-04-10 (Actual); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: Post-Traumatic Stress Disorder; Prevention; Propranolol; Psychophysiology
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Propranolol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Propranolol (Experimental): Following the occurrence of an acute psychologically traumatic event, an initial dose of short-acting propranolol 40 mg orally then one hour later, long-acting propranolol 60 mg capsule orally on Day 1 followed by a 19-day course of long-acting propranolol starting with 120 mg every morning and evening for 10 days, and then tapering to 120 mg in the morning and 60 mg in the evening for 3 days, then 60 mg in the morning and 60 mg the evening for 3 days, then 60 mg in the morning for 3 days.
  Interventions: Drug: Propranolol
- Placebo (Placebo Comparator): Following the occurrence of an acute psychologically traumatic event, an initial dose of placebo-matching short-acting propranolol 40 mg orally then one hour later, placebo-matching long-acting propranolol 60 mg capsule orally on Day 1 followed by a 19-day course of placebo-matching long-acting propranolol starting with 120 mg every morning and evening for 10 days, and then tapering to 120 mg in the morning and 60 mg in the evening for 3 days, then 60 mg in the morning and 60 mg the evening for 3 days, then 60 mg in the morning for 3 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Propranolol — Propranolol short-acting or long-acting capsule
  Other Names: Inderal
  Arms: Propranolol
Drug: Placebo — Placebo-matching propranolol short-acting or long-acting capsule
  Arms: Placebo

SUMMARY:
This study will assess the effectiveness of taking propranolol soon after a traumatizing incident in reducing the incidence and severity of posttraumatic stress disorder in acutely traumatized individuals.

DETAILED DESCRIPTION:
Posttraumatic Stress Disorder (PTSD) is a psychiatric disorder that can occur following exposure to a traumatic event in which grave physical harm occurred or was threatened. PTSD is marked by clear biological changes as well as psychological symptoms. Many people with PTSD repeatedly relive the trauma in the form of flashback episodes, memories, nightmares, or frightening thoughts. This study will assess the effect of post-trauma propranolol on reducing the incidence and severity of PTSD. The study will also evaluate propranolol's effectiveness as a preventive measure against subsequent PTSD symptoms.

Participants in this double-blind study will be recruited upon admission to the Massachusetts General Hospital Emergency Department after exposure to a psychologically traumatic event. Baseline psychometric and psychobiologic measurements will be collected. Within 6 hours following the traumatic event, participants will be randomly assigned to receive either 40 mg of short-acting propranolol or placebo and 60 mg of either long-acting propranolol or placebo. For the next 10 days, participants will receive 120 mg of either long-acting propranolol or placebo twice daily. A 9-day medication tapering will follow. Participants will undergo psychophysiologic, psychodiagnostic, and psychometric testing for PTSD 1 and 3 months following the traumatic event.

ELIGIBILITY:
Inclusion Criteria:

* Experienced an acute psychological traumatic event
* Heart rate of 80 beats per minute (bpm) or greater
* Understands English

Exclusion Criteria:

* Traumatic event that occurred more than four hours before arrival to emergency department
* Physical injury that may affect safe participation (e.g., head injury)
* Systolic blood pressure less than 100 mm Hg
* Medical or surgical condition that poses a risk of shock
* Medical condition that may affect the safe administration of propranolol
* Previous adverse reaction to, or non-compliance with, a beta-blocker
* Current use of medication that may react badly with propranolol
* Elevated saliva alcohol level
* Presence of salivary opiates, marijuana, cocaine, or amphetamines
* Pregnant or breastfeeding
* Traumatic event reflecting ongoing victimization
* Psychiatric condition that may affect safe participation
* Unwilling or unable to commute to Boston for research visits
* Attending physician in emergency department does not advise participation

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2004-09 (Actual); Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger K. Pitman, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts

REFERENCES:
- [Result] Hoge EA, Worthington JJ, Nagurney JT, Chang Y, Kay EB, Feterowski CM, Katzman AR, Goetz JM, Rosasco ML, Lasko NB, Zusman RM, Pollack MH, Orr SP, Pitman RK. Effect of acute posttrauma propranolol on PTSD outcome and physiological responses during script-driven imagery. CNS Neurosci Ther. 2012 Jan;18(1):21-7. doi: 10.1111/j.1755-5949.2010.00227.x. Epub 2011 Jan 10. PMID 22070357
- [Derived] Bertolini F, Robertson L, Bisson JI, Meader N, Churchill R, Ostuzzi G, Stein DJ, Williams T, Barbui C. Early pharmacological interventions for prevention of post-traumatic stress disorder (PTSD) in individuals experiencing acute traumatic stress symptoms. Cochrane Database Syst Rev. 2024 May 20;5(5):CD013613. doi: 10.1002/14651858.CD013613.pub2. PMID 38767196
- [Derived] Bertolini F, Robertson L, Bisson JI, Meader N, Churchill R, Ostuzzi G, Stein DJ, Williams T, Barbui C. Early pharmacological interventions for universal prevention of post-traumatic stress disorder (PTSD). Cochrane Database Syst Rev. 2022 Feb 10;2(2):CD013443. doi: 10.1002/14651858.CD013443.pub2. PMID 35141873

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who experienced a qualifying acute psychological trauma were randomized to receive up to 240 mg/day of propranolol or placebo.
Period: Overall Study
Arm/Group | Placebo | Propranolol
Started | 21 | 22
Completed | 20 | 21
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants with data available for analysis. 1 participant in each arm dropped out prior to analysis and are excluded.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Propranolol | Total
Number analyzed (Participants) | 20 | 21 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 21 | 41
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.8 (9.4) | 33.3 (11.0) | 33.6 (10.2)
Sex/Gender, Customized [Number; unit: participants]
  Female | 7 | 10 | 17
  Male | 13 | 11 | 24
Region of Enrollment [Number; unit: participants]
  United States | 20 | 21 | 43

OUTCOME MEASURES:

1. Primary Outcome: Physiological Posterior Probability of Posttraumatic Stress Disorder (PTSD) as Determined From Psychophysiologic Responses During Script-Driven Mental Imagery at Month 1
Description: The posterior probability of developing PTSD was determined for each participant from a composite of psychophysiological responses during script-driven mental imagery of traumatic events (two exemplars) that included assessments of heart rate response in beats per minute, skin conductance response in microSiemens, and corrugator and left lateral frontalis facial muscle electromyogram (EMG) responses in microVolts. Responses for the two traumatic scripts were averaged and square-root transformed for analysis. Responses during personal traumatic imagery of previously studied individuals with and without current PTSD were used to calculate each participant's posterior probability of being classified as PTSD.
Time Frame: Month 1
Population: All randomized participants with data available for analysis at Month 1. Data were missing in 2 placebo and 2 propranolol participants.
Measure: Mean (Standard Deviation); unit: percent probability
Arm/Group | Placebo | Propranolol
Number analyzed (Participants) | 18 | 19
percent probability | 40.7 (17.0) | 33.7 (10.2)
Statistical Analysis 1: Comparison: Placebo vs Propranolol; Test type: Superiority; Mean Difference (Final Values) = 7.0, 95% CI 2-sided [-2.7 to 16.7] — Placebo-Propranolol

2. Secondary Outcome: Clinician-Administered PTSD Scale (CAPS) Total Score
Description: The clinician evaluated the overall frequency and intensity/severity of the participant's PTSD symptoms using the CAPS. 17 Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM-IV) PTSD symptoms were assessed using a 5-point scale for intensity where 0=none to 4=extreme and a 5-point scale for frequency where 0=never to 4=most or all of the time. The intensity score and the frequency scores were added together for a total possible score of 0 (best) to 136 (worst).
Time Frame: Months 1 and 3
Population: All randomized participants with CAPS data available for analysis at the given time-point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Propranolol
Number analyzed (Participants) | 20 | 21
score on a scale
  Month 1 | 28.5 (27.1) | 28.5 (21.5)
  Month 3: number analyzed (Participants) | 17 | 17
  Month 3 | 19.0 (25.8) | 21.2 (26.1)
Statistical Analysis 1: Comparison: Placebo vs Propranolol; CAPS Total Score at Month 1; Test type: Superiority; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-15.5 to 15.3] — Placebo-Propranolol
Statistical Analysis 2: Comparison: Placebo vs Propranolol; CAPS Total Score at Month 3; Test type: Superiority; Mean Difference (Final Values) = -2.2, 95% CI 2-sided [-20.3 to 16.0]

3. Primary Outcome: Physiological Posterior Probability of PTSD as Determined From Psychophysiologic Responses During Script-Driven Mental Imagery at Month 3
Description: as for outcome 1
Time Frame: Month 3
Population: All randomized participants with data available for analysis at Month 3. Data were missing in 6 placebo and 5 propranolol participants.
Measure: Mean (Standard Deviation); unit: percent probability
Arm/Group | Placebo | Propranolol
Number analyzed (Participants) | 14 | 16
percent probability | 34.9 (13.1) | 32.0 (5.8)
Statistical Analysis 1: Comparison: Placebo vs Propranolol; Test type: Superiority; Mean Difference (Final Values) = 2.9, 95% CI 2-sided [-4.8 to 10.7] — Placebo-Propranolol

ADVERSE EVENTS:
Time Frame: Up to 3 Months
Description: All randomized participants with data available for analysis. 1 participant in each arm dropped out prior to analysis and are excluded.
Arm/Group | Placebo | Propranolol
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/21
Other Adverse Events (participants affected / at risk) | 0/20 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No